CLINICAL TRIAL: NCT06871995
Title: Efficacy, Safety and Limitations of Spinal Block When Used for All Infants Under 3 Months of Age Scheduled for Lower Abdominal Surgery
Brief Title: Efficacy, Safety and Limitations of Spinal Block for All Infants Under 3 Months
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD234/2024
Record Dates: First submitted 2025-02-21; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: spinal block in infants less than 3 months of age undergoing lower abdominal surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- one arm All Infants Under 3 Months of Age receiving Spinal Block (Experimental): All Infants Under 3 Months of Age Scheduled for Lower Abdominal Surgery
  Interventions: Procedure: spinal block

INTERVENTIONS:
Procedure: spinal block — All patients will receive spinal anesthesia via midline approach with patients in sitting position established by assistant under complete aseptic conditions. A subcutaneous bleb using Lidocaine 1% through the needle of an insulin syringe followed by minor skin scratch to will help avoiding possible intrathecal dermoid implantation . A lumbar puncture will be performed in L4-L5 or L5- S1 interspace using 25-G 25-mm pencil-point spinal needle . Depth of epidural space is anticipated at 0.1 mm/kg . After getting free flow of cerebrospinal fluid (CSF) hyperbaric bupivacaine (0.5%) in a dose of 0.5 mg/kg (0.1 ml/kg) will be slowly injected in the subarachnoid space . The end of the injection will be taken as time zero for further data recording.

SUMMARY:
Spinal anesthesia (SA) has been shown to be a viable alternative to general anesthesia (GA) for infants and children for a variety of surgical procedures. SA serves to avoid some of the potential risks of GA including the need for airway manipulation, hemodynamic instability, postoperative apnea, and exposure to medications that may cause neurotoxicity .SA allows the prevention and reduction of perioperative complications even if its duration is an important limiting factor. Because of this limitation, short surgery is the most indicated under SA . Premature infants and neurologically impaired children account for the majority of spinal anesthetics used today .

This study evaluates the effectiveness, safety and limitations of spinal anesthesia when used for all infants under 3 months undergoing lower abdominal surgery at Ain Shams University Hospitals.

DETAILED DESCRIPTION:
Patients will be carefully examined 24 hours (h) to the procedure and every case will be assessed individually concerning its eligibility for spinal anesthesia under the supervision of a senior pediatric anesthesiologist. History taking and clinical examination along with the necessary laboratory tests . Standard blood test is cbc and we will use it a routine before surgery. About 1 ml blood is needed as a sample.

Counseling the parents or the legal guardian regarding every aspect of the procedure and obtaining their informed written consent.

All patients will be fasting from formula milk for 6 hours, breast milk for 4 hours and clear fluid for 1 h before anesthesia . No overnight premedication will be given.

After the establishment of intravenous access, all patients will be given crystalloid solution (Ringer's solution or Normal Saline) of 10 ml/kg over 30 minutes started with the application of monitors. Heart rate, blood pressure, oxygen saturation. Blood glucose level is measured.

The monitors will be connected and pulse oximetry (SPO2) baseline non-invasive blood pressure (NIBP), heart rate (HR), and electrocardiogram (ECG tracings) will be obtained. Fluid bolus of 5 ml/kg will be used for any intraoperative hypotension. Atropine 50µ/kg will be given intravenously if HR dropped > 20% of baseline reading . Intraoperative blood loss will be replaced by 3 times volume with the same crystalloid .blood glucose level is measured after injection then every 30 minutes till end of surgery .

All patients will receive spinal anesthesia via midline approach with patients in sitting position established by assistant under complete aseptic conditions. A subcutaneous bleb using Lidocaine 1% through the needle of an insulin syringe followed by minor skin scratch to will help avoiding possible intrathecal dermoid implantation . A lumbar puncture will be performed in L4-L5 or L5- S1 interspace using 25-G 25-mm pencil-point spinal needle . Depth of epidural space is anticipated at 0.1 mm/kg . After getting free flow of cerebrospinal fluid (CSF) hyperbaric bupivacaine (0.5%) in a dose of 0.5 mg/kg (0.1 ml/kg) will be slowly injected in the subarachnoid space . The end of the injection will be taken as time zero for further data recording.

Since the Bromage score is not assessable among this pediatric population, the success of the spinal anesthesia is estimated and based on the presence of profound motor block (unable to move feet, knees and legs) in the lower extremities and the absence of a skin prick response using toothed forceps at the appropriate dermatome level. If these signs will not confirmed after 5 min, general anesthesia will be performed . All of these cases will be registered as spinal block failure Then pacifier dipped with sugar water will be offered to the baby.

Throughout the operation, the effect of the spinal anesthesia will be monitored till return of spontaneous movement or response to surgical stimulus then sevoflurane mask will be applied and surgery continues either mask or even intubation then mean time of conversion to general anesthesia will be recorded and registered as spinal block failure.

Complications from SA:

Hypotension is defined as a more than 20%decrease in mean blood pressure from baseline. (Mean blood pressure =post conceptual age in weeks ).

Bradycardia is defined as a heart rate less than 120 b/min or HR dropped > 20% of baseline reading) Apnea is defined as a sustained respiratory pause of 15 s or longer or less than15s if accompanied by oxygen saturation (SpO2) less than 90% or bradycardia. Hypoxemia is defined as oxygen saturation below 90% .

High spinal block is defined as apnea after spinal injection without sedative drugs and/or motor block of the upper extremities and no response to hand finger pinprick All this complications will be monitored intra and postoperatively and managed accordingly.

All patients will be admitted postoperative for 12 hours in the hospital. Post operative cbc also a routine blood test will be done .The conductors of this study will record the degree of motor block and pain. The pain control will be measured using the Face, Legs, Activity, Crying, and Controllability (FLACC) pain score (0-10 score range) . The FLACC score will be evaluated and recorded during the first 12h immediately postoperative and at 2, 4, 6, 12 hours postoperatively. The time of giving analgesia (intravenous paracetamol 15 mg/kg) will be recorded when the FLACC score exceeds 4, with a maximum of four doses per day, and total paracetamol consumption will be recorded . It is given that pain medications will be given when the FLACC score exceeds 4 at assessment or in between of the allotted time interval.

ELIGIBILITY:
Inclusion Criteria

* Age under 3 months.
* Physical status: American Society of Anesthesiologists I - II.
* Elective lower abdominal surgeries such as: hernia, hydrocele, undescended testis

Exclusion Criteria:

* Patient's parents or legal guardian refusing to do this specific procedure.
* Coagulopathy, use of anti-coagulant or antiplatelet therapy.
* Infection at the site of injection.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
the success rate of spinal block in abdominal surgeries in infants under 3 months of age. | during the surgery
  Success rate = (no of total patients - no of all converted general anesthesia patients) divided by no of total cases%.

SECONDARY OUTCOMES:
Duration of spinal block in minutes | during the surgery
  Duration of spinal block
Number of attempts | during the surgery
  Number of attempts till success
Depth of insertion of the spinal needle | during the surgery
  from skin to subarachnoid space
Blood glucose level | every 30 minutes till end of surgery
  sample to measure blood glucose
Determine the incidence of complications | after spinal block to end of surgery
  1. Apnea that will be considered as high spinal block
  2. Hypotension (a more than 20% decrease in systolic blood pressure from baseline.)
  3. Bradycardia (a heart rate less than120 /min or HR dropped > 20% of baseline reading)
  4. Hypoxemia (oxygen saturation below 90%) .

CONTACTS AND LOCATIONS:
Overall Officials: hany mo Elzahaby, prof, Study Director — Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt